CLINICAL TRIAL: NCT02485964
Title: A Pilot Study to Assess the Immunogenicity of Candidate PSA Peptides for a Prostate Cancer Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 204374
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2021-09-10 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: Vaccine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Draw Only (Other): One time blood draw at time of consent; No treatment
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — One time blood draw at time of consent. Blood will be stored until all subjects have been enrolled and then the enzyme-linked immunospot (ELISPOT) assay will be done to measure the antigen-specific interferon secretion.

SUMMARY:
To measure antigen-specific interferon-secretion by enzyme-linked immunospot (ELISPOT) assay, which measures antigen-specific interferon-secretion.

DETAILED DESCRIPTION:
The goal of this project is to collect information in regards to the immunogenicity of PSA peptides in order to develop a novel therapeutic vaccine. This vaccine will consist of prostate specific antigen (PSA) peptide and Candida skin test reagent. Candida has recently been shown to be a promising new vaccine adjuvant for promoting T-cell responses. It can induce interleukin-12 (promotes T-cell response) secretion by Langerhans cells, the main antigen presenting cells in skin. In a Phase I clinical trial treating women with biopsy-proven high-grade squamous intraepithelial lesions (HSILs), precursors of cervical cancer, a combination of human papillomavirus peptides with Candida was demonstrated to be safe, to induce immune responses to human papillomavirus, and to promote T-helper type 1 (Th-1) response (promotes cellmediated immunity) in vaccine recipients.

For treating prostate cancer, PSA is an ideal antigen as it is expressed in prostate cancer but not in any other organs. The characteristics of peptides that can effectively be used in therapeutic vaccines are their solubility in a single solution, immunogenicity in terms of containing large number of T-cell epitopes (so the vaccine can be used for all patients and not just a few that express certain Human Leukocyte Antigen (HLA) tissue types), and ability to mature Langerhans cells which in turn promotes T-cell activity.

In this protocol the investigators focus on the immunogenicity of candidate peptides.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented diagnosis of prostate cancer
* 18 years of age or older
* Signed informed consent form approved by the University of Arkansas for Medical Sciences (UAMS) Institutional Review Board (IRB)

Exclusion Criteria:

* Subjects must have no other current malignancies.
* Subjects with prior history at any time of any basal or squamous skin cancer are eligible, provided they are disease-free at the time of registration.
* Subjects with other malignancies are eligible if they have been continuously disease free for ≥ 5 years prior to the time of registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Arnaoutakis, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Draw Only
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blood Draw Only
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 72 [64 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antigen-specific Interferon- Secretion as Measured by Enzyme-linked Immunospot (ELISPOT) Assay
Description: The spots formed by interferon-gamma-secreting T-cells will be counted with an automated ELISPOT analyzer (AID ELISPOT Classic Reader; Autoimmune Diagnostika GmbH, Strassberg, Germany). The average spot-forming units (SFU) per antigen will be calculated. A response will be considered positive when the average SFU in wells with a given peptide was at least twice that of the average SFU in the no-peptide control wells.
Time Frame: At time of consent
Measure: Number; unit: participants
Arm/Group | Blood Draw Only
Number analyzed (Participants) | 10
participants | 4

ADVERSE EVENTS:
Time Frame: at time of enrollment (1 day)
Arm/Group | Blood Draw Only
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02485964/Prot_SAP_000.pdf